CLINICAL TRIAL: NCT06027658
Title: Psychotherapeutic Care of Women Victims of Sexual Violence, Longitudinal Comparative Study and Therapeutic Evaluation of a Dance As Therapy Program
Brief Title: Validation of a Dance As Therapy Program in Co-facilitation
Acronym: VaDDanC
Status: Completed | Type: Observational
Sponsor: University of Franche-Comté (Other)
Collaborators: University of Lorraine (Other); University of Roehampton (Other); LOBA association (Unknown)
Responsible Party: Principal Investigator, Crystal Tomaszewski, Principal Investigator, University of Franche-Comté
Other Study IDs: CERUBFC-2021-11-09-035
Record Dates: First submitted 2023-08-01; First posted 2023-09-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Trauma, Psychological; Depression, Anxiety; Stress; Body Image; Quality of Life; Social Relationship; Attachment Disorder
Keywords: Sexual violence; Trauma; Psychotherapy; Dance as therapy; Longitudinal study; Attachment; Mentalization
MeSH Terms: conditions — Psychological Trauma; Depression; Anxiety Disorders; Wounds and Injuries | interventions — Recreation Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non participants: Individuals receiving the standard support for victims of sexual violence (e.g. medical, social, and legal assistance, individual psychotherapy)
- Participants: Individuals receiving the RECREATION program in addition to standard support for victims of sexual violence
  Interventions: Behavioral: RECREATION therapy
- Long term participants: Individual receiving the RECREATION program for at least a month
  Interventions: Behavioral: RECREATION therapy
- Professionals: Professionals associated with long term participants, working with them for standard support

INTERVENTIONS:
Behavioral: RECREATION therapy — Dance as therapy program with speech and movement co-therapy via body activity.
  Groups: Long term participants; Participants

SUMMARY:
The objective is to validate a psychotherapeutic group protocol of dance as therapy created by LOBA association with a comparative non-randomized study.

DETAILED DESCRIPTION:
This present research is a prospective longitudinal monocentric comparative study of an alternative, non-pharmacological therapy. It is a controlled, non-randomized, and experimental study in which half of the participants benefit from an additional program with speech and movement co-therapy via body activity, and the other half only benefit from standard support (e.g. medical, social, and legal assistance, individual psychotherapy).

The effect of this program will be examined across three dimensions:

* A clinical trial of N=80 participants to compare symptom improvement between individuals receiving the standard support for victims of sexual violence (N=40) and those receiving, in addition, the RECREATION program (N=40).
* A longitudinal evaluation of physiological conditions, psychological traits, and social well-being of RECREATION workshop attendees (N=10) versus victims not participating in said workshops (N=10).
* A qualitative analysis of interviews with program participants and their associated professionals (data saturation sample size).

ELIGIBILITY:
Inclusion Criteria:

* French-speaking
* Woman
* Over 18 years old
* Victim of sexual violence

Exclusion Criteria:

* Non-French-speaking person,
* Under 18 years old
* Not woman
* Not victim of sexual violence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migration-affected adult women (over 18 years old) victims of sexual violence, mostly born in Subsaharian African Countries.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Rate of participants presenting an improvement in PCLS scores at 6 months | 6 months period between January 2022 and April 2024
  Posttraumatic stress disorder checklist (PCLS) scores range from 0 to 85; a higher score means a worse outcome.
Rate of participants presenting an improvement in DASS-21 scores at 6 months | 6 months period between January 2022 and April 2024
  Depression, Anxiety, and Stress Scale in 21 (DASS-21) items scores range from 0 to 63; a higher score means a worse outcome.
Rate of participants presenting an improvement in QSCPGS scores at 6 months | 6 months period between January 2022 and April 2024
  Body satisfaction and global self-perception questionnaire (QSCPGS) scores range from -100 to +100; a higher score means a better outcome
Rate of participants presenting an improvement in SF-36 scores at 6 months | 6 months period between January 2022 and April 2024
  Short Form Health Survey in 36 items (SF-36) scores range from 0 to 100; a higher score means a better outcome
Rate of participants presenting an improvement in SSQ6 scores at 6 months | 6 months period between January 2022 and April 2024
  Social Support Questionnaire in 6 items (SSQ6) scores range from 0 to 54 for the availability subscale and from 6 to 36 for the satisfaction subscale. For both subscales, a higher score means a better outcome
Rate of participants presenting a change in RSQ score at 6 months | 6 months period between January 2022 and April 2024
  Relationship Scales Questionnaire (RSQ) scores give an attachment profile, attachment strategies and a self and other model.
Rate of participants presenting an improvement in RFQ8 score at 6 months | 6 months period between January 2022 and April 2024
  Reflexive Functioning Questionnaire in 8 items (RFQ8) scores range from 0 to 18; a higher score means a worse outcome.
Number of participants presenting an improvement in Rorschach protocol at 1 year | A year between April 2022 and December 2023
  Rorschach protocols are interpreted both qualitatively and quantitatively (psychogram). This outcome focuses on trauma symptomatology.
Number of participants presenting an improvement in AAI scores at 1 year | A year between April 2022 and December 2023
  Adult Attachment Interview (AAI) scores range from 0 to 90; a higher score means a better outcome.
Number of identical themes in participants' and professionals' semi-structured interviews | One interview per person between September 2022 and March 2023
  Number of identical themes in participants' and professionals' semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Rose-Angélique Belot, Study Director — Université de Franche-Comté, Fr; Crystal Tomaszewski, Principal Investigator — Université de Franche-Comté, Université de Lorraine, LOBA, Fr; Aziz Essadek, Study Director — Université de Lorraine, Fr; Christophe Clesse, Study Director — University of Roehampton, UK
Locations (1):
- LOBA, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tomaszewski, C., Essadek, A., Onumba-Bessonnet, H., Clesse, C. et Belot, R.-A. (2024). Violences sexuelles, traumatismes et mentalisation, Etude de la dynamique psychique à partir du cas Hélène. L'Evolution Psychiatrique. https://doi.org/10.1016/j.evopsy.2024.06.002
- [Background] Tomaszewski C, Belot RA, Essadek A, Onumba-Bessonnet H, Clesse C. Impact of dance therapy on adults with psychological trauma: a systematic review. Eur J Psychotraumatol. 2023;14(2):2225152. doi: 10.1080/20008066.2023.2225152. PMID 37427835